CLINICAL TRIAL: NCT01934400
Title: Osteoporosis and Fall Prevention Education With High Risk Population Telephone Follow up Study
Brief Title: Osteoporosis and Fall Prevention Education
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201303003RINC
Record Dates: First submitted 2013-08-26; First posted 2013-09-04 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; fall prevention; high risk population
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: The study is to increasing osteoporosis awareness with fracture risk assessments and management as well as fall prevention among elderly in northern region of Taiwan.

Method: Six community osteoporosis and fall prevention educational programme will be held at northern region of Taiwan. A questionnaires design including demographic variables , FRAX variables, nutritional variables and osteoporosis and fall knowledge variables as well.The pretest-posttest method was used to analyse the effect on education.

Expected outcomes : (1)Fall prevention educational programme will hold in northern region of Taiwan at different communities in order to increasing osteoporosis awareness with fracture risk assessment tool, establishing fall knowledges among elderly and some fall prevention skills.(2)Elderly with 10-year probability of major osteoporotic fracture risk who more than 20% and 10-year probability of hip fracture risk who more than 3% will identify as high risk of osteoporosis. (3) To estimate number of cases who identified as high risk will recommend for BMD measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between the ages of 40 to 90.
2. Adults who been fractures prior to assessment.
3. Adults who have ability, well conscious to complete the questionnaires.

Exclusion Criteria:

1.Adults who have treatment currently will not include in this study.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who attending the fall prevention educational programme.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Measurement of effects of fall prevention education. | 6-months
  The primary outcomes is to determine the effects after investigaor given the fall prevention education. The pretest-posttest method was used to analyse the effect on education.

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, MD,PHD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan